CLINICAL TRIAL: NCT03748225
Title: The Fami-Life Study: Protocol of a Prospective Multicenter Observational Mixed Study of Psychological Consequences of Grieving Families in French Palliative Care Units on the Behalf of the F.R.I.P.C Research Network
Brief Title: Incidence and Risk Factors of Prolonged Grief in Palliative Care Units
Acronym: FAMI-LIFE
Status: Completed | Type: Observational
Sponsor: Hôpital Franco-Britannique-Fondation Cognacq-Jay (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Principal Investigator, Maité Garrouste-Orgeas, MD, Director, head of clinical research, principal investigator, medical doctor, Hôpital Franco-Britannique-Fondation Cognacq-Jay
Other Study IDs: IHFB-002
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-01

CONDITIONS: Bereaved Families

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the incidence and risk factors of prolonged grief in family members of patients died in French palliative care units and to explore experience of bereaved families to build a scientifically valid management prevention program.

DETAILED DESCRIPTION:
There is hardly knowledge on how bereavement is treated in palliative care patient's relatives. The field of bereavement needs studies that validate the theoretical underpinning of the research area. This study will depict the grieving process of individuals having lost a relative in palliative care in France. Having baseline data of incidence of prolonged grief, risk factors of relative's prolonged grief and identification of risk factors associated with the management of end-of-life issues in palliative care will contribute to target interventions that should help decrease bereaved families burden.

The investigator designed a quantitative study to assess the psychological effect of families after the death of the patient in palliative care unit and a qualitative study to examine the grieving prolonged process.

ELIGIBILITY:
Inclusion Criteria:

* Families of adult patients hospitalized more than 72 hours in a palliative care unit for end-of-life care.
* Eligibility of end-of-life cares are defined after the first evaluation by the palliative care physician.

Exclusion Criteria:

* Patients with less than 72 hours of life-expectancy
* Patients or families who refused the study
* Patients or families included in a study using the same questionnaires
* Patients without families visiting them in the first 24 hours after admission
* Patients not hospitalized for end-of-life issues
* Families not fluent in French
* Deaf or mute families

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participating palliative care units belong to the French Society of Palliative Care (SFAP) and are selected using the list of the different French units on their website. An invitation of participation is sent to the clinical responsible of each unit.
  The participating units belong to university, community and private hospitals.
Sampling Method: Probability Sample
Enrollment: 609 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Incidence of prolonged grief in bereaved family members | 6 months after patient's death in palliative care unit
  Inventory Grief Disorder > 25
Risk factors of prolonged grief in bereaved family members | 6 months after patient's death in palliative care unit
  Hierarchical logistic regression models with a random effect center after selection of variables by univariate analysis then introduced in a multivariate analysis

SECONDARY OUTCOMES:
Post traumatic stress disorder in bereaved family members | 6 months after patient's death in palliative care unit
  Impact of event Scale-revised > 22
Anxiety and depression symptoms in bereaved family members | 6 months after patient's death in palliative care unit
  Hospital anxiety and depression scale ≥ 8
Anxiety and depression symptoms in family members | Between between day 3 and day 5 after patient admission in the palliative care unit
  Hospital anxiety and depression scale ≥ 8
Report of the families' grief experience in those who have signs of prolonged grief according to the Inventory of Complicated Grief questionnaire with a score > 25 | Between 6 and 12 months after the patient' death.
  Interpretative Phenomenological Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Timsit, MD, PhD, Study Chair — INSERM 1137, IAME, Paris Diderot University, Paris
Locations (1):
- French British Institute, Levallois-Perret, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fasse L, Flahault C, Bredart A, Dolbeault S, Sultan S. Describing and understanding depression in spouses of cancer patients in palliative phase. Psychooncology. 2015 Sep;24(9):1131-7. doi: 10.1002/pon.3777. Epub 2015 Feb 24. PMID 25707938
- [Result] Kentish-Barnes N, Chaize M, Seegers V, Legriel S, Cariou A, Jaber S, Lefrant JY, Floccard B, Renault A, Vinatier I, Mathonnet A, Reuter D, Guisset O, Cohen-Solal Z, Cracco C, Seguin A, Durand-Gasselin J, Eon B, Thirion M, Rigaud JP, Philippon-Jouve B, Argaud L, Chouquer R, Adda M, Dedrie C, Georges H, Lebas E, Rolin N, Bollaert PE, Lecuyer L, Viquesnel G, Leone M, Chalumeau-Lemoine L, Garrouste M, Schlemmer B, Chevret S, Falissard B, Azoulay E. Complicated grief after death of a relative in the intensive care unit. Eur Respir J. 2015 May;45(5):1341-52. doi: 10.1183/09031936.00160014. Epub 2015 Jan 22. PMID 25614168
- [Result] Flahault C, Dolbeault S, Sankey C, Fasse L. Understanding grief in children who have lost a parent with cancer: How do they give meaning to this experience? Results of an interpretative phenomenological analysis. Death Stud. 2018 Sep;42(8):483-490. doi: 10.1080/07481187.2017.1383951. Epub 2018 Jan 24. PMID 29173097
- [Result] Fasse L, Sultan S, Flahault C, Mackinnon CJ, Dolbeault S, Bredart A. How do researchers conceive of spousal grief after cancer? A systematic review of models used by researchers to study spousal grief in the cancer context. Psychooncology. 2014 Feb;23(2):131-42. doi: 10.1002/pon.3412. Epub 2013 Sep 30. PMID 24115499
- [Derived] Garrouste-Orgeas M, Flahault C, Poulain E, Evin A, Guirimand F, Fossez-Diaz V, Perruchio S, Verlaine C, Vanbesien A, Kaczmarek W, Birkui de Francqueville L, De Lariviere E, Bouquet G, Copel L, Verliac V, Marche V, Mathias C, Gracia D, Mhalla A, Michonneau-Gandon V, Poupardin C, Touzet L, Ranchou G, Guastella V, Richard B, Bienfait F, Sonrier M, Michel D, Ruckly S, Bailly S, Timsit JF. The Fami-life study: protocol of a prospective observational multicenter mixed study of psychological consequences of grieving relatives in French palliative care units on behalf of the family research in palliative care (F.R.I.P.C research network). BMC Palliat Care. 2019 Dec 9;18(1):111. doi: 10.1186/s12904-019-0496-4. PMID 31818281